CLINICAL TRIAL: NCT06555484
Title: Acute Effects of Supplemental Oxygen on Memory in Healthy Older Adults: a Double-Blind Within-Subject Crossover Study
Brief Title: Acute Effects of Supplemental Oxygen on Memory Testing in Healthy Adult Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: INO-06
Record Dates: First submitted 2024-07-27; First posted 2024-08-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Cognition
Keywords: Oxygen Concentrator; Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Intervention Model Description: Acute effects of oxygen on memory testing in healthy adult volunteers
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Air First (Other): All study participants, completing memory tests while breathing either supplemental oxygen followed by air, or breathing air followed oxygen.
  Interventions: Device: Cross Over Assignment Supplemental Oxygen and Supplemental Air
- Oxygen First (Other): All study participants, completing memory tests while breathing either supplemental oxygen followed by air, or breathing air followed oxygen.
  Interventions: Device: Cross Over Assignment Supplemental Oxygen and Supplemental Air

INTERVENTIONS:
Device: Cross Over Assignment Supplemental Oxygen and Supplemental Air — Subjects repeatedly complete memory tests, either first while breathing supplemental oxygen or first while breathing "supplemental air" (in an order randomly assigned).

SUMMARY:
Forty healthy adults (i.e., not recruited with respect to any particular diagnosis) are each alternately provided with supplemental oxygen and air via nasal cannula at about 6 Liters per Minute (LPM), while completing memory tests.

DETAILED DESCRIPTION:
Prior studies have reported that supplemental oxygen can confer acute benefits to cognition. Here, the investigators seek to replicate/extend such findings by assessing whether such benefits can be seen using an Inogen oxygen concentrator with subjects with an average age around 65 years old. The investigators include a standard measure of cognition previously reported to be sensitive to supplemental oxygen (2-back test) and a novel, in-development adaptation of a memory test for medical-related content (Medical icons spatial test).

ELIGIBILITY:
Inclusion Criteria:

Subjects are intended to represent "healthy adults." Patients will include a mix of self-reported gender and ethnic/racial identification.

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Adult (aged 22+)

Exclusion Criteria:

* Patients who self-report diagnosis of respiratory-related conditions will be excluded.
* Subjects with a known polyvinyl chloride (PVC) allergy will be excluded, due to potential use of a standard, PVC-based cannula in the study.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
2 back Memory test performance | At baseline and 5 mins post-intervention exposure
  # correct on 2-back test
Memory test performance | At baseline and 5 mins post-intervention exposure
  New Medical Icons Spatial Test

CONTACTS AND LOCATIONS:
Overall Officials: Marc Egeth, Principal Investigator — Inogen Inc.
Locations (1):
- Two Liberty Place, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi MH, Kim HJ, Kim JH, Kim HS, Choi JS, Yi JH, Tack GR, Chung YS, Son I, Chung SC. Correlation between cognitive ability measured by response time of 1-back task and changes of SpO2 by supplying three different levels of oxygen in the elderly. Geriatr Gerontol Int. 2013 Apr;13(2):384-7. doi: 10.1111/j.1447-0594.2012.00911.x. Epub 2012 Jul 23. PMID 22817401
- [Background] Chung SC, Kwon JH, Lee HW, Tack GR, Lee B, Yi JH, Lee SY. Effects of high concentration oxygen administration on n-back task performance and physiological signals. Physiol Meas. 2007 Apr;28(4):389-96. doi: 10.1088/0967-3334/28/4/005. Epub 2007 Mar 7. PMID 17395994
- [Background] McMorris T, Hale BJ, Barwood M, Costello J, Corbett J. Effect of acute hypoxia on cognition: A systematic review and meta-regression analysis. Neurosci Biobehav Rev. 2017 Mar;74(Pt A):225-232. doi: 10.1016/j.neubiorev.2017.01.019. Epub 2017 Jan 19. PMID 28111267
- [Background] Sohn JH, Chung SC, Jang EH. 30% oxygen inhalation enhances cognitive performance through robust activation in the brain. J Physiol Anthropol Appl Human Sci. 2005 Jan;24(1):51-3. doi: 10.2114/jpa.24.51. PMID 15684544
- [Background] Shaw DM, Bloomfield PM, Gant N. The effect of acute normobaric hyperoxia on cognition: A systematic review, meta-analysis and meta-regression. Physiol Behav. 2023 Aug 1;267:114208. doi: 10.1016/j.physbeh.2023.114208. Epub 2023 Apr 29. PMID 37121344
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/37121344/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/15684544/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/28111267/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/22817401/